CLINICAL TRIAL: NCT06198790
Title: Postoperative Anemia After Bariatric Surgery
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Yuntao Nie, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: CJBariatric005
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Anemia; Bariatric Surgery Candidate
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the real incidence of short and long-term anemia after bariatric surgery, and explore the risk factors.

DETAILED DESCRIPTION:
This study aims to investigate the real incidence of short and long-term anemia after bariatric surgery and explore the risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo sleeve gastrectomy or Roux-en-Y gastric bypass
* Aged between 16 and 70 years
* Patients who is not diagnosed as anemia at baseline

Exclusion Criteria:

* Patients who have anemia at baseline

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients without anemia at baseline who will undergo bariatric surgery will be included.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of anemia after 1, 3, 5, 10 years | 10 years
  Incidence of anemia after 1, 3, 5, 10 years

SECONDARY OUTCOMES:
Incidence of anemia-related nutrient deficiencies | 10 years
  Incidence of folate, ferritin, vitamin B12, and iron deficiencies
Hazard ratios for the risk factors of postoperative anemia | 10 years
  Hazard ratios for the risk factors of postoperative anemia will be calculated by Cox regression model.

CONTACTS AND LOCATIONS:
Overall Officials: Yuntao Nie, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- Yuntao Nie, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Data should be accessed with the permission of the principal investigator.